CLINICAL TRIAL: NCT02092142
Title: Evaluation of the Safety and Immunogenicity of Q Fever Vaccine, Phase I, Inactivated, Dried, NDBR 105, in Subjects at Risk of Exposure to Coxiella Burnetii
Brief Title: Safety and Immunogenicity of Q Fever Vaccine
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: US Army Medical Research Institute of Infectious Diseases (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: S-11-19; FY13-02 (Other: MRMC)
Record Dates: First submitted 2014-03-17; First posted 2014-03-20 (Estimated); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Q Fever
Keywords: Q fever; Coxiella burnetii
MeSH Terms: conditions — Q Fever | interventions — Clinical Trials, Phase I as Topic; Desiccation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vaccinated (Experimental): The vaccine will be administered subcutaneously in the upper outer aspect of the arm (triceps area) with 0.5 mL Q fever Vaccine, Phase I, Inactivated, Dried, NDBR 105 (which equals 30 μg)
  Interventions: Biological: Q fever Vaccine

INTERVENTIONS:
Biological: Q fever Vaccine — Subcutaneous 0.5 mL Q fever Vaccine, Phase I, Inactivated, Dried, NDBR 105
  Other Names: Q fever Vaccine, Phase I, Inactivated, Dried, NDBR 105

SUMMARY:
The purpose of this study is to evaluate the safety of Q Fever Vaccine, Phase I, Inactivated, Dried, NDBR 105 and collect data on incidence of occupational Q fever infection in vaccinated personnel.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old.
* Females of childbearing potential must agree to have a urine pregnancy test on the same day before receipt of skin test AND vaccine. (Exception: documented hysterectomy or ≥ 3 years of menopause.) The results must be negative. Females must agree to not become pregnant for 3 months after receipt of the skin test or vaccination.
* Considered at risk for exposure to C burnetii and who have submitted a Request for Investigational New Drug (IND) Vaccines for the Q Fever vaccine.
* Sign and date the approved informed consent document and Health Insurance Portability and Accountability Act (HIPAA) Authorization.
* Have on their charts:

  * Up-to-date medical history (including concomitant medications)
  * Physical examination and laboratory tests within 1 year
  * Previous chest x-ray and electrocardiogram
* Be medically cleared for participation by an investigator. Examinations or tests may be repeated at the discretion of the enrolling physician.
* Willing to return for all follow-up visits.
* Agree to report any adverse events (AEs) that may or may not be associated with administration of the test article for at least 28 days after vaccination and agree to report all serious adverse events (for example, resulting in hospitalization) for the duration of the subject's participation in the study (6 months).
* Agree to defer blood, bone marrow, and organ donation for 1 year after receipt of skin test antigen and/or vaccine.

Exclusion Criteria:

* Prior history of Q fever disease or vaccination.
* Clinically significant abnormal lab results (including evidence of hepatitis C, hepatitis B carrier state) or elevated liver function tests (two times the normal range or at the discretion of the principal investigator).
* Personal history of an immunodeficiency or current treatment with an oral or intravenous immunosuppressive medication.
* Confirmed HIV infection.
* Heart valve disease: prosthetic heart valve or clinically significant heart murmur. (If a murmur is detected on examination, an echocardiogram may be obtained or subject may be referred to a cardiologist to determine clinical significance.)
* Aneurysm/vascular graft.
* Joint prosthesis.
* History of chronic fatigue syndrome (or positive by chronic fatigue syndrome (CFS) Questionnaire criteria).
* Positive pregnancy test or breast-feeding female.
* Any known allergies to components of the vaccine:

  * Formalin
  * Eggs or chicken products
* Administration of another vaccine or investigational product within 28 days of skin test and subsequent Q fever vaccination.
* Any unresolved AE resulting from a previous immunization.
* Transplant recipients, subjects with cancer, and those with chronic kidney disease.
* A medical condition that, in the judgment of the principal investigator, would impact subject safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-02; Primary Completion 2019-02 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Change in Immunogenicity | Day 28, Day 56, or 6 months
  Immune response will be evaluated for per protocol subjects to determine the percentage of subjects who experience a ≥ fourfold rise in immunofluorescence assay (IFA) antibody titer after vaccination. Immunoglobulin M (IgM) at Day 28 or Day 56, or immunoglobulin G (IgG) at 6 months.
Percentage of subjects with symptoms following Q fever vaccination | 6 months
Percentage of subjects with erythema following Q fever vaccination along with severity and association with vaccination | 6 months
Percentage of subjects with induration following Q fever vaccination along with severity and association with vaccination | 6 months
Percentage of subjects with each AE, system organ class of AE, severity, and association with vaccination | 6 months
Percentage of subjects with symptoms following Q fever skin test antigen | 6 months
Percentage of subjects with erythema following Q fever skin test antigen along with severity and association with skin test antigen | 6 months
Percentage of subjects with induration following Q fever skin test antigen along with severity and association with skin test antigen | 6 months
Percentage of subjects with each AE, system organ class of AE, severity, and association with skin test antigen | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Goldberg, MD, Principal Investigator — Special Immunizations Program, USAMRIID
Locations (1):
- Special Immunizations Program, Division of Medicine, USAMRIID, Fort Deterick, Maryland, United States